CLINICAL TRIAL: NCT05245110
Title: Tri-Service General Hospital, National Defense Medical Center
Brief Title: Effectiveness of Tele-exercise Training on Cardiorespiratory Fitness in Patients With Cardiometabolic Multimorbidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, CHIA-HUEI LIN, PhD, Associate Professor and Deputy Director of Nursing Department, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSGHIRB: 1-106-05-107
Record Dates: First submitted 2022-01-29; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Heart Diseases; Type 2 Diabetes; Metabolic Syndrome; Coronary Artery Disease; Heart Failure
Keywords: exercise; physical activity; cardiorespiratory fitness
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus, Type 2; Metabolic Syndrome; Coronary Artery Disease; Heart Failure; Motor Activity

STUDY DESIGN:
Intervention Model Description: A parallel-group randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Eligible participants were invited to data collection including sociodemographic characteristics and outcome measures in a local medical centre at baseline and 12 weeks by a separate research nurse, blinded to the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): received a tele-exercise training program
  Interventions: Behavioral: tele-exercise training
- control group (No Intervention): usual care only

INTERVENTIONS:
Behavioral: tele-exercise training — a 12-week tele-exercise training program
  Arms: experimental group

SUMMARY:
This trial aimed to assess whether assumed increase in physical activity after tele-exercise training can improve cardiorespiratory fitness of patients with cardiometabolic multimorbidity.

DETAILED DESCRIPTION:
A parallel-group randomized controlled trial was conducted. Eligible patients with cardiometabolic multimorbidity were randomized 1:1 to either experimental group (EG, received a tele-exercise training program) or control group (CG, usual care only). The intervention encompassed tele-exercise training program (30 min/session, 3 sessions/week) and weekly remote monitoring for maintenance of exercise. Physical activity and cardiorespiratory fitness were assessed at baseline and 12 weeks. Generalized estimating equations were used to examine the intervention effects via the interaction of time and group.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnoses of cardiometabolic multimorbidity, defined as the presence of two or more cardiometabolic conditions (i.e., hypertension, type 2 diabetes, hyperlipidaemia, heart disease, metabolic syndrome, or gout)
* Aged 18-80 years
* Able to speak and understand Mandarin
* Able to walk without assistance
* Had mobile phones and could easily access the Internet

Exclusion Criteria:

* Not match the diagnosis of cardiometabolic multimorbidity; and a history of arrhythmia, cancer, end-stage renal disease with dialysis, being diagnosed with mental illness, recent stroke within 6 months
* Not able to speak and understand Mandarin
* Not able to walk independently or inability to participate due to comorbid neurological, musculoskeletal conditions that produce moderate-to-severe physical disability
* Did not have mobile phones or could not access the internet at home and whenever necessary

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline physical activity amount at 12 weeks | 12 weeks
  weekly amount of physical activity using the well-validated and reliable Taiwan version of 7-item International Physical Activity Questionnaire to measure. The scores of International Physical Activity Questionnaire expressed as "MET-minutes/week". Higher score indicates higher physical activity amounts
Changes from baseline VO2 peak (ml/kg/min) at 12 weeks | 12 weeks
  VO2 peak (ml/kg/min), detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline workload (Watts)at 12 weeks | 12 weeks
  Workload (Watts), detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline anaerobic threshold at 12 weeks | 12 weeks
  anaerobic threshold, detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline O2 pulse (ml/beat) at 12 weeks | 12 weeks
  O2 pulse (ml/beat), detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline One-min heart rate recovery (beat) at 12 weeks | 12 weeks
  One-min heart rate recovery (beat), detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline Two-min heart rate recovery (beat) at 12 weeks | 12 weeks
  Two-min heart rate recovery (beat), detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline resting heart rate (bpm) at 12 weeks | 12 weeks
  Resting heart rate (bpm) obtained using electronic BP monitor devices (Terumo, ESP2000)
Changes from baseline Resting Systolic Blood Pressure (mmHg) at 12 weeks | 12 weeks
  Resting Systolic Blood Pressure (mmHg) obtained using electronic BP monitor devices (Terumo, ESP2000)
Changes from baseline Resting Diastolic Blood Pressure (mmHg) at 12 weeks | 12 weeks
  Resting Diastolic Blood Pressure (mmHg), obtained using electronic BP monitor devices (Terumo, ESP2000)
Changes from baseline forced vital capacity (L/min) at 12 weeks | 12 weeks
  forced vital capacity (L/min), detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes form baseline forced expiratory volume in one second (L/min) at 12 weeks | 12 weeks
  forced expiratory volume in one second (L/min), detected during graded exercise testing, performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline FEV1/FVC (%) at 12 weeks | 12 weeks
  FEV1/FVC (%) detected during graded exercise testing, , performed using a motorized ergometer (Corival, Lode, Netherlands) with a standardized ramp protocol by increasing the resistance (10 watt per minute) at a consistent speed of 60 revolutions per minute.
Changes from baseline Ejection fraction (%) at 12 weeks | Baseline and 12 weeks
  Ejection fraction (%) data were collected through chart review
Changes from baseline BNP at 12 weeks | 12 weeks
  BNP through blood analysis
Changes from baseline Health-related quality of life at 12 weeks | 12 weeks
  Health-related quality of life useing the reliable and valid Taiwan version of Medical Outcomes Study Short-Form 36 to measure. Scores ranged from 0 to 100, with higher scores indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Huei Lin, PhD, Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Chia-Huei Lin, Taipei, Hawaii, Taiwan